CLINICAL TRIAL: NCT05680532
Title: The Improvement of Black Raspberry in Obese and Mild AZ Patients Infected With H. Pylori
Acronym: BR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Chin Kun Wang, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CS2-21103
Record Dates: First submitted 2022-12-07; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Alzheimer Disease; H Pylori Infection
Keywords: black raspberry; Alzheimer's patients; H pylori; Inflammatory cytokines; Antioxidant
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BR group (Experimental): Experimental group AZ subjects were requested to take 50 g of BR powder dissolved in 240 ml of water for 4 weeks.
  Interventions: Dietary Supplement: Black raspberry
- Placebo group (Placebo Comparator): Placebo group AZ subjects were requested to take 50 g of dextrin powder dissolved in 240 ml of water for 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Black raspberry — Experimental group subjects were requested to take 50 g of Black Raspberry powder for 4 weeks.
  Arms: BR group
Other: Placebo — Placebo group subjects were requested to take 50 g of dextrin for 4 weeks.
  Arms: Placebo group

SUMMARY:
The current study was designed to check the impact of black raspberry (BR) on obese and mild Alzheimers (AZ) patients infected with Helicobacter pylori (H pylori). Through checking various parameters including anthropometric, antioxidants, and CDR.

DETAILED DESCRIPTION:
The current study was designed to check the impact of black raspberry (BR) on obese and mild Alzheimers (AZ) patients infected with Helicobacter pylori (H pylori).

Preclinical studies (In vitro model) were conducted using 3T3-L1 adipocyte cells to check the anti-adhesion activity of BR.

For the clinical trial, a total of 21 obese mild AZ patients were recruited and separated into 2 groups: Experimental (BR group) and Placebo group.

Experimental group and Placebo group subjects were requested to take either 50 g of BR or 50 g of dextrin respectively for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≧ 27, Waist circumference: men ≧ 90cm, women ≧ 80cm,
* Body fat: male ≧ 25%, female ≧ 30%,
* UBT 13C test value> 10‰ (H. pylori (+)),
* CDR (clinical dementia rating) = 0.5

Exclusion Criteria:

* BMI< 27
* Severe chronic diseases (liver disease, cardiovascular disease, kidney disease)
* Alcohol abuse
* Smoking habit
* Taking berry-related supplementation or any known allergies related to berries.
* Subjects with prior history of H. pylori infection were treated with triple therapy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Glycemic indices | 8 weeks
  No significant changes in any of the glycemic indices
Anthropometric parameters | 8 weeks
  BMI were significantly altered

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Kun Wang, Ph.D, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tandoro Y, Chiu HF, Tan CL, Hsieh MH, Huang YW, Yu J, Wang LS, Chan CH, Wang CK. Black raspberry supplementation on overweight and Helicobacter pylori infected mild dementia patients a pilot study. NPJ Sci Food. 2025 Feb 12;9(1):9. doi: 10.1038/s41538-024-00356-w. PMID 39939643